CLINICAL TRIAL: NCT00191009
Title: Atomoxetine Augmentation of Cholinesterase Inhibitor Therapy in Patients With Alzheimer's Disease
Brief Title: Adding Atomoxetine To Standard Medication Treatment In Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7951; B4Z-MC-LYCG
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: atomoxetine hydrochloride
Drug: placebo

SUMMARY:
This study will compare atomoxetine to placebo when taken with current standard Alzheimer's Disease medications. The treatment will take approximately 6 months and it is hypothesized atomoxetine will significantly improve cognitive performance as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents with Alzheimer's Disease based on clinical history.
* Patient must have a Mini Mental Status Score between 10 and 26.
* Patient must have a reliable caregiver in frequent or daily contact with the patient.
* Patient must be currently treated with and on a stable dose of a standard Alzheimer's drug treatment for at least 3 months.

Exclusion Criteria:

* Patients who are receiving pharmacologic treatments (other than a cholinesterase inhibitor or memantine) for Alzheimer's Disease.
* Patients who have a history in the past 5 years or any current evidence of major psychiatric illness.
* Patients who have narrow angle glaucoma.
* Patients who are experiencing clinically significant urinary hesitancy or retention as assessed by a physician.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124
Dates: Start 2003-10; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To see if Alzheimer's patients receiving a stable dose of an Alzheimer's drug randomly assigned to atomoxetine for approximately 6 months will have cognitive performance improved as measured by the Alzheimer's Disease Assessment Scale - Cognitive

SECONDARY OUTCOMES:
To see if patients taking an Alzheimer's medication plus atomoxetine for approximately 6 months will be superior to an Alzheimer's medication alone as assessed by the Clinician's Interview-Based Impression of Change (CIBIC+) score.
To see if patients taking an Alzheimer's medication plus atomoxetine will display less comorbid psychological symptoms, such as depression, as assessed by the Neuropsychiatric Inventory (NPI). Patients will receive the NPI once before randomization
To see if current Alzheimer's medications plus atomoxetine compared to Alzheimer's medications plus placebo is better at preserving or slowing cognitive decline as measured by the Alzheimer's Disease Cooperative Study Inventory - Activities of
To show that current Alzheimer's drugs can be taken with atomoxetine without significant side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Wichita Falls, Texas

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com